CLINICAL TRIAL: NCT00086047
Title: Randomized Clinical Trial in Juvenile Fibromyalgia
Brief Title: Coping Skills Training for Adolescents With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR050028 (NIH); R01AR050028 (NIH)
Record Dates: First submitted 2004-06-22; First posted 2004-06-23 (Estimated); Results first posted 2013-11-06 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: Fibromyalgia
Keywords: Juvenile Fibromyalgia Syndrome; JPFS; Fibromyalgia; Chronic Pain; Pediatric Pain; Juvenile Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Cognitive Behavioral Therapy; Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping Skills (Experimental): Patients will receive 8 weeks of behavioral training in pain coping strategies
  Interventions: Behavioral: Coping Skills Training
- Education (Active Comparator): Patient will receive 8 weekly sessions of education about fibromyalgia syndrome.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Coping Skills Training — 8 weekly sessions of behavioral treatment
  Other Names: cognitive-behavioral therapy
  Arms: Coping Skills
Behavioral: Education — 8 weekly sessions of fibromyalgia education
  Arms: Education

SUMMARY:
Juvenile fibromyalgia is a chronic pain condition that can cause considerable suffering and difficulty in an adolescent's day-to-day activities. The purpose of this study is to determine whether coping skills training, when combined with usual medical care, can reduce pain and disability in adolescents with fibromyalgia.

Study hypotheses: 1) Adolescents who receive coping skills training combined with their usual medical care will show significantly greater reductions in functional disability, pain, and depressive symptoms at the end of the acute treatment phase than adolescents who receive fibromyalgia education with their usual medical care. 2) Adolescents who receive coping skills training with their usual medical care will show significantly lower levels of functional disability, pain, and depressive symptoms at the end of a six-month maintenance phase than adolescents who receive fibromyalgia education with their usual medical care.

DETAILED DESCRIPTION:
Juvenile Primary Fibromyalgia Syndrome (JPFS) is a debilitating chronic pain condition that occurs in adolescence and is characterized by persistent pain, multiple tender points, sleep difficulty, and fatigue. The cause of JPFS is unknown and there is no known cure. Children and adolescents with JPFS have difficulty with daily functioning, miss a great deal of school, and experience increased emotional distress compared to their peers. Fibromyalgia syndrome appears to be resistant to treatment in adulthood, so early behavioral treatment for JPFS with long-term beneficial effects would be useful. This study will evaluate the efficacy of coping skills training (CST) when combined with usual medical care in reducing functional disability, pain intensity, and depressive symptoms in adolescents with JPFS. This study will also determine whether improvements can be sustained long-term.

This study will last 34 weeks. Participants will be recruited from three pediatric rheumatology clinics. Patients will be randomly assigned to one of two groups: CST plus usual medical care or education plus usual medical care. There will be 6 medical visits, spaced 4 to 5 weeks apart. In addition, patients will attend 8 individual sessions of CST or education over the first 8 weeks of the study. CST sessions will include training in cognitive-behavioral techniques of pain management for the adolescent and behavioral management techniques for their parents. Education sessions will include education on fibromyalgia and discussion about lifestyle issues, but no training in pain management procedures.

Patients will be evaluated at Week 9 and will be followed for an additional 6-month maintenance phase. During this maintenance phase, adolescents will continue to receive their usual medical care and will attend 2 additional sessions of CST or education. There will be one final evaluation at the end of the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of JPFS based upon widespread pain for over 3 months, at least 5 tender points, and associated features such as sleep difficulty, fatigue, and abdominal discomfort
* Average pain intensity greater than 4 on the Visual Analog Scale
* Functional disability score greater than 7
* Stable medications for 8 weeks prior to study entry

Exclusion Criteria:

* Other chronic rheumatic diseases, such as juvenile rheumatoid arthritis or lupus
* Significant developmental delay or impairments, such as autism, cerebral palsy, or mental retardation
* Present or lifetime psychiatric diagnosis that meets DSM-IV criteria for panic disorder, bipolar disorder, major depressive disorder, or psychosis
* Opioid medications are disallowed when used on an ongoing basis for treatment of fibromyalgia pain

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 114 (Actual)
Dates: Start 2004-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susmita Kashikar-Zuck, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (3):
- United States (3):
  - Kosair Charities Pediatric Center, Louisville, Kentucky
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Division of Pediatrics, Cleveland, Ohio

REFERENCES:
- [Result] Kashikar-Zuck S, Ting TV, Arnold LM, Bean J, Powers SW, Graham TB, Passo MH, Schikler KN, Hashkes PJ, Spalding S, Lynch-Jordan AM, Banez G, Richards MM, Lovell DJ. Cognitive behavioral therapy for the treatment of juvenile fibromyalgia: a multisite, single-blind, randomized, controlled clinical trial. Arthritis Rheum. 2012 Jan;64(1):297-305. doi: 10.1002/art.30644. PMID 22108765
- [Derived] Joffe NE, Lynch-Jordan A, Ting TV, Arnold LM, Hashkes PJ, Lovell DJ, Passo MH, Powers SW, Schikler KN, Kashikar-Zuck S. Utility of the PedsQL rheumatology module as an outcome measure in juvenile fibromyalgia. Arthritis Care Res (Hoboken). 2013 Nov;65(11):1820-7. doi: 10.1002/acr.22045. PMID 23686969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with juvenile fibromyalgia (ages 11-18 years)were recruited from four pediatric rheumatology clinics in the Midwestern United States.
Pre-assignment Details: Patients were screened to determine eligibility for the study. if they met eligibility criteria, they were enrolled in the study and immediately randomized to one of the treatment arms.
Period: Overall Study
Arm/Group | Coping Skills | Education
Started | 57 | 57
Completed | 50 | 50
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 7 | 6
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coping Skills | Education | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 57 | 57 | 114
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.8) | 14.9 (1.7) | 15.0 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 105
  Male | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  United States | 57 | 57 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change in FDI (Functional Disability Inventory) Scores at End of Study
Description: Functional disability score is measured by the Functional Disability Inventory (FDI)which assesses ability to engage in usual physical, social and recreational activities. Scores range from 0=no disability to 60 = extreme disability and and are interpreted as No/Mild disability (0-12); Moderate Disability (13-29) and Severe Disability (30-60)
Time Frame: Baseline and 6 months (end of study)
Population: Intent to treat analysis
Measure: Mean (95% Confidence Interval); unit: units on a 0-60 scale
Groups:
- Coping Skills Training: Consists of training in pain management skills using cognitive-behavioral therapy techniques
- Fibromyalgia Education: Consists of education about fibromyalgia and its management
Arm/Group | Coping Skills Training | Fibromyalgia Education
Number analyzed (Participants) | 57 | 55
units on a 0-60 scale
  Baseline FDI Score | 21.4 (9.4) [18.9 to 23.9] | 19.2 (8.2) [17.0 to 21.3]
  End of Study FDI Score | 13.4 (8.9) [10.9 to 15.9] | 17.0 (10.5) [14.0 to 19.9]
Statistical Analysis 1: Comparison: Coping Skills Training vs Fibromyalgia Education; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; Mean Difference (Final Values) = 5.39, 95% CI 2-sided [1.57 to 9.22], Standard Deviation 8.8

2. Secondary Outcome: Pain Intensity
Time Frame: 9 weeks and 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Depressive Symptoms
Time Frame: 9 weeks and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: ITT population
Arm/Group | Coping Skills | Education
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/55
Other Adverse Events (participants affected / at risk) | 0/57 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No